CLINICAL TRIAL: NCT02811926
Title: Incidence and Risk Factors of Parastomal Bulging in Patients With Ileostomy or Colostomy: a Register-based Study
Brief Title: Incidence and Risk Factors of Parastomal Bulging in Patients With Ileostomy or Colostomy
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Rune Martens Andersen, PhD fellow, Rigshospitalet, Denmark
Other Study IDs: 15018151
Record Dates: First submitted 2016-05-30; First posted 2016-06-23 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Colostomy; Ileostomy - Stoma; Enterostomy
Keywords: parastomal bulging; peristomal bulging; ileostomy; colostomy; enterostomy; incidence; risk factor

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ileostomy or colostomy: Patients with a ileostomy or colostomy in the Capital Region of Denmark

SUMMARY:
The purpose of this study is to use routinely-collected health data from registers to examine the incidence of parastomal bulging (PB) at different time points in the first year after surgery for ileostomy or colostomy. Additionally, the purpose is to investigate risk factors for development of PB.

DETAILED DESCRIPTION:
Parastomal bulging (PB) in patients with ileostomy and colostomy in the Capital Region of Denmark up to one year after surgery is the primary outcome in this study. The investigators will use a register-based study design to evaluate routinely-collected health data from the Danish Stoma Database Capital Region (DSDCR). Incidence of PB one year post surgery and at different points of follow-up during the first year will be investigated using survival analysis. Potential risk factors will be investigated controlling for potential confounders. In order to include relevant variables on lifestyle, comorbidity, and physical status, data from the DSDCR will be linked to data from the Danish Anaesthesia Database.

ELIGIBILITY:
Inclusion Criteria:

* Subject is registered in the Danish Stoma Database Capital Region
* Is registered as having either ileostomy, jejunostomy, sigmoidostomy, or transversostomy

Exclusion Criteria:

* Patients with urostomy or unknown stoma type

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with an ileostomy or colostomy in the Danish Stoma Database Capital Region
Sampling Method: Non-Probability Sample
Enrollment: 5019 (Actual)
Dates: Start 2016-07; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with the incidence of parastomal bulging | Up to 1 year after primary surgery
  Parastomal bulging evaluated by stoma care nurses through symptoms, visual inspection, and stomal exploration. Parastomal bulging is evaluated at scheduled visits at stoma care clinics on postoperative days 30, 90, 180, and 365, and at any additional visits inbetween.

IPD SHARING:
Plan to Share IPD: No